CLINICAL TRIAL: NCT06524557
Title: Department of Ultrasonic Medicine, The First Affiliated Hospital of Air Force Medical University
Brief Title: Exploration of Noninvasive Differential Diagnosis of Benign and Malignant Liver Tumors
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-20180101-3
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Liver Tumor
Keywords: liver tumors; benign; malignant; Differential diagnosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with chronic liver disease: patients with hepatitis B virus, hepatitis C virus and other chronic liver disease.
  Interventions: Diagnostic Test: with chronic liver disease
- without chronic liver disease: patients without hepatitis B virus, hepatitis C virus and other chronic liver disease.

INTERVENTIONS:
Diagnostic Test: with chronic liver disease — patients with hepatitis B virus，hepatitis C virus, or other chronic liver disease
  Groups: with chronic liver disease

SUMMARY:
To explore an effective noninvasive method for differential diagnosis of liver tumors.

DETAILED DESCRIPTION:
A retrospective study was performed to assess the performance of certain ultrasound-based parameters, in distinguishing benign from malignant with liver biopsy as the gold standard. Demographic data, clinical information and serological data were obtained from participants who were retrospectively enrolled. Receiver operating characteristic (ROC) curve analysis was conducted, including calculation of the optimal area under the ROC curve (AUC), to assess the performance of these measures in distinguishing between benign and malignant in patients with or without chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

(1) age 18-70 years; (2) liver examination performed for all patients prior to US-guided liver biopsy or surgery; (3) tumor can be visualized in conventional US; (4) largest tumor sectional area saved in DICOM format for use in later analyses; (5) a histopathological diagnosis made either from US-guided liver biopsy or surgical resection; (6) suitable routine clinical and US data obtained within 7 days of the histopathological diagnosis.

Exclusion Criteria:

(1) unavailable pathological diagnosis; (2) liver metastatic tumors; (3) poor quality US images; and (4) a past history of surgical resection, percutaneous local ablation, radiation, transarterial and systemic therapies or liver transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 200 patients whose pathological diagnoses were confirmed by US-guided liver biopsy or surgery and who underwent preoperative conventional US between January 2018 and November 2025 were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The differential diagnosis of liver tumors | 2018.01-2025.12
  Multimodal ultrasound is of great value in the differential diagnosis of liver tumors

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Huihui, M.M., Study Chair — Department of Ultrasonic Medicine, The First Affiliated Hospital of Air Force Medical University
Locations (1):
- Xijing Hosptial, Xi'an, Xi'an, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou H, Sang L, Sun Y, Gong X, Zhang J, Liu L, Wei J, Jiao W, Yu M. Performance of Ultrasonography-Based Fractal Parameters in Distinguishing Hepatocellular Carcinoma From Intrahepatic Cholangiocarcinoma. Ultrason Imaging. 2025 Jul;47(3-4):115-124. doi: 10.1177/01617346251330257. Epub 2025 Apr 15. PMID 40231713